CLINICAL TRIAL: NCT07027826
Title: Use of the Esophageal String Test as a Diagnostic Screening Tool for Eosinophilic Esophagitis Among Africans With Dysphagia in Mali and the United States
Brief Title: The Esophageal String Test as a Diagnostic Screening Tool for Eosinophilic Esophagitis Among Africans With Dysphagia in Mali and the United States
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10002313; 002313-I
Record Dates: First submitted 2025-06-18; First posted 2025-06-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12-05

CONDITIONS: Dysphagia; Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis; Dysphagia; Esophageal string test
MeSH Terms: conditions — Deglutition Disorders; Eosinophilic Esophagitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Esophageal string test (Experimental): The esophageal string test is a minimally invasive procedure used to collect esophageal secretions for diagnostic analysis.
  Interventions: Device: Esophageal string test

INTERVENTIONS:
Device: Esophageal string test — The esophageal string test consists of a gelatin or cellulose capsule containing a nylon string. The capsule dissolves allowing the nylon string to absorb esophageal secretions which can be analyzed for various inflammatory mediators.

SUMMARY:
Background:

Eosinophilic esophagitis (EoE) is a disease that causes inflammation in the esophagus. The esophagus is the tube that moves food from the mouth to the stomach. Diagnosing EoE currently requires a specialized tool called an endoscope. The esophageal string test (EST) is another test; the EST collects fluid from the upper digestive tract. An EST is simpler and cheaper than an endoscopy. Researchers want to know if an EST can diagnose EoE.

Objective:

To test if the EST can diagnose EoE in people who have trouble swallowing.

Eligibility:

Adults aged 18 to 65 years with trouble swallowing. They must have been born in Africa and be of African descent.

Design:

Participants will be screened. They will give blood, stool, urine, and skin swab samples. They will complete surveys about their medical history, diet, symptoms, and home environment. They will bring a sample of their drinking water for testing.

Participants will have an EST. They will swallow a pill capsule that contains a nylon string. One end of the string will be taped to their cheek. The string will unravel down the esophagus and into the stomach. It will be pulled out after 1 hour. Fluids that soaked into the string will be tested.

At a different visit, participants will have an endoscopic exam. An endoscope is a flexible tube that is inserted down the mouth; it can be used to take tissue samples from the esophagus, stomach, and small intestine.

Participants will have a final visit in person, online, or by phone. They will take a survey and talk about their test results.

DETAILED DESCRIPTION:
Study Description:

Eligible participants will be enrolled to assess the performance and accuracy of the 1-hour esophageal string test (EST) as a diagnostic screening tool for eosinophilic esophagitis (EoE). Consenting participants in the U.S. (n=30) and Mali (n=30) undergoing clinically indicated esophagogastroduodenoscopy (EGD) will have an EST performed prior to the procedure. Clinical data, including medical history and laboratory test results, will be captured on a case report form. Symptoms will also be assessed using validated patient reporting outcome measures: the Brief Esophageal Dysphagia Questionnaire (BEDQ) and Patient-Reported Outcomes Measurement Information System (PROMIS-GI and -57). Dietary, sociodemographic, and environmental histories will be obtained by validated questionnaires. Blood, urine, stool, and skin swab/tape strip samples will be obtained for additional biomarker studies.

Participants will be screened for intestinal helminth infections by stool polymerase chain reaction (PCR). Tissue samples obtained during EGD will be assessed for Helicobacter pylori by histopathology. Esophageal biopsy samples and remaining EST eluents will be allocated for investigational studies. Air and water samples will be collected from areas within the participants community and analyzed to determine potential correlation with elevated levels of environmental pollutants. The hypothesis of this study is that the 1-hour EST will provide a preliminary estimate of EoE prevalence among Africans and African immigrants presenting with dysphagia.

Primary Objective:

-Assess the accuracy of the 1-hour EST as a diagnostic screening tool for EoE among African-born individuals presenting with dysphagia in the U.S. and Mali.

Secondary Objective:

-Determine the frequency of EoE among African-born individuals presenting with dysphagia in the U.S. and Mali.

Primary Endpoint(s):

* Sensitivity, as estimated by the proportion of positive EST-obtained EoE-Score(TM) results out of those diagnosed with EoE by the gold standard of esophageal biopsy.
* Specificity, as estimated by the proportion of negative EST-obtained EoE-Score(TM) results out of those diagnosed with EoE by the gold standard of esophageal biopsy.

Secondary Endpoints:

-Proportion of EoE cases diagnosed in each cohort.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Able to provide informed consent.
2. Aged 18 to 65 years.
3. Born in the African continent and of African ancestry.
4. Exhibiting symptoms of dysphagia and/or prior history of food impaction.
5. Undergoing clinically indicated endoscopy at the NIH Clinical Center or Centre Hospitalier Universitaire Gabriel Toure and willing to provide research samples and data.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Recent steroid use (systemic or swallowed/topical corticosteroid) within 4 weeks prior to endoscopy.
2. Recent use of dupilumab (Dupixent) within the last 6 months.
3. Recent use of other biologic medications (within either 6 months or 5 half-lives, whichever is longer). Examples of biologic medications include:

3a. mepolizumab (Nucala)

3b. reslizumab (Cinqair, Cinqaero)

3c. benralizumab (Fasenra)

3d. cendakimab

3e. tezepelumab (Tezspire)

3f. barzolvolimab

4. Individuals suffering from a bleeding diathesis (e.g., hemophilia, severe thrombocytopenia).

5. Current use of anticoagulant medications.

6. Pregnancy.

7. Treatment with another investigational drug or other investigational intervention within 6 months or 5 half-lives whichever is longer.

8. Individuals with a known history of any of the following:

8a. eosinophilic esophagitis

8b. esophageal stricture unable to be passed with an upper endoscope

8c. esophageal cancer

8d. esophageal motility disorder (e.g., achalasia)

8e. esophageal varices

8f. esophageal or gastric surgery including fundoplication

8g. neurologic cause of dysphagia (e.g., stroke, Parkinson s disease, etc.)

8h. allergy to gelatin

8i. inability to swallow pills

9. Any condition that, in the investigator s opinion, places the individual at undue risk by participating in the study.

Co-enrollment guidelines: Co-enrollment in other trials is restricted, other than enrollment on observational studies. Consideration for co-enrollment in trials evaluating the use of a licensed medication will require the approval of the principal investigator in consultation with the medical monitor. Study staff should be notified of co-enrollment on any other protocol as it may require the approval of the principal investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the esophageal string test to detect Eosinophilic Esophagitis. | End of study
  Assess the accuracy of the 1-hour EST as a diagnostic screening tool for EoE in populations with limited access to subspecialty care. Sensitivity and specificity provide a measure of accuracy when compared to the diagnostic gold standard.

SECONDARY OUTCOMES:
Proportion of Eosinophilic Esophagitis cases diagnosed in each cohort. | End of study
  Determine the frequency of EoE among African-born individuals presenting with dysphagia in the U.S. and Mali. Allows for the comparison of diagnostic rates across different groups, providing insights into the prevalence.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Constantine, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States
- Gabriel Toure University Hospital Center, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002313-I.html